CLINICAL TRIAL: NCT04867486
Title: Reliability and Validity of Urdu Version of the Dynamic Gait Index in Pakistani Geriatric Population
Brief Title: Urdu Version of the Dynamic Gait Index: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00262
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Balance
Keywords: Dynamic gait index; balance; reliability; validity; geriatric population

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, Investigators will observe the reliability and validity of dynamic gait index in Urdu language in Pakistani geriatric population with balance impairments.

DETAILED DESCRIPTION:
The aim of study is to translate and culturally adapt DGI into Urdu language and secondly to investigate the reliability and validity of DGI in geriatrics Pakistani population.This study will be cross sectional survey in which convenience sampling technique will be used to enroll participants as per pre-defined criteria.

The results of study will help to know the validity and reliability of DGI in Urdu version with balance impairments in geriatric population.The reliability of the scale will be checked through internal consistency and test-retest methods. Internal consistency will be analyzed with Cronbach's alpha value.Test-retest reliability will be assessed using an intraclass correlation coefficient with 60 patients

ELIGIBILITY:
Inclusion Criteria:

* Age at least 65 years
* Ability to walk a minimum of 6m with or without a walking Aid
* One or more falls in the last year or
* Observed balance impairment evaluated subjectively by a physical therapist during the initial training session (Time Up and Go test, Morse Fall Scale)

Exclusion Criteria:

* Inability to understand or follow the instructions of the DGI
* Experience with the DGI in the last 6 months
* Acute illness or fracture in the lower extremities or knee/hip replacement within the last 3 months.

Ages: 65 Years to 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly people, especially those of the advanced ages, suffer from coexistent disorders, many of which are chronically degenerative, falls and gait disorders are common issues. About one-third of all elderly people aged 65 as well as above fall at least once a year. Injury, physical impairments, morbidity, cognitive side effects, and even disability are all linked to fall because equilibrium and postural control are essential for the everyday work.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | 1st day
  The Dynamic Gait Index tests the participant's ability to maintain balance while walking under different dynamic conditions and at the same time to react to different task requirements. An order scale with four points in the range from 0 to 3. "0" indicates the lowest functional level and "3" the highest functional level. The score of 19 predicts falls in the elderly and> 22 out of 24 in safe ambulances
Dynamic Gait Index | 2nd day
  The Dynamic Gait Index tests the participant's ability to maintain balance while walking under different dynamic conditions and at the same time to react to different task requirements. An order scale with four points in the range from 0 to 3. "0" indicates the lowest functional level and "3" the highest functional level. The score of 19 predicts falls in the elderly and> 22 out of 24 in safe ambulances falls is the dynamic gait index.Each object is marked at a scale of 0 to 3, 3 with standard and 0 showing led to problems DGI's 24 is the highest result possible

SECONDARY OUTCOMES:
Berg Balance Scale | 1st day
  The Berg balance scale is an objective assessment of balance performance based on 14 items common to everyday activities. it is a 14-item scale that rates 0 (unable to perform) to 4 (normal performance) for each item. The total score is 56 points. Higher score higher balance ability.
Time Up and Go Test | 1st day
  Time Up and Go Test is used determine fall risk and measure the progress of balance, sit to stand and walking, Cut of scores indicating risk of falls by Population Community Dwelling adults - 13.5 in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No